CLINICAL TRIAL: NCT06449599
Title: Outcomes of Rhomboid Intercostal Plane Block on Local Anesthesia in Cardiac Implantable Electronic Device Implantation: A Randomized Controlled Clinical Trial
Brief Title: RIB for Perioperative Analgesia in CIED Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kerem Erkalp, MD, Prof, proffessor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 015
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Postoperative Pain; Arrhythmias, Cardiac
Keywords: rhomboid intercostal plane block,; postoperative analgesia; cardiac electrophysiology; cardiac implantable electronic devices; arrhythmia; satisfaction
MeSH Terms: conditions — Pain, Postoperative; Arrhythmias, Cardiac; Personal Satisfaction | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The RIB procedure for the intervention group will be performed in a separate room 60 minutes prior to the patient's transfer to the cardiac electrophysiology laboratory, as described in the methodology section. When the patient arrives at the electrophysiology lab, the cardiologist performing the CIED implantation is not informed whether RIB has been administered beforehand. However, due to the nature of the study, patients are not blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- block group (Active Comparator): local anesthesia will be applied to surgical field as a part of the routine procedure and additionally rhomboid intercostal plane block will be applied
  Interventions: Device: ultrasound
- control group (Sham Comparator): only local anesthesia will be applied to surgical field as a part of the routine procedure.
  Interventions: Procedure: parenteral local anesthesia

INTERVENTIONS:
Device: ultrasound — Local anesthesia 400 mg(20ml) prilocaine 2% to surgical field and additionally ultrasound-guided RIB with 0,25% bupivacaine 20 ml will be applied to the patients who will be inserted cardiac implantable electronic devices An additional 100 mg of prilocaine will be administered as the first-line rescue treatment if the intraoperative NRS-11 score was ≥4.If the patient has an NRS-11 score of ≥4 again during the procedure,100 mg of prilocaine will be administered again as the second rescue treatment.
  In the postoperative follow-up of the patients,1 g of paracetamol will be administered IV as an infusion for 20 minutes as the first rescue treatment if the patients have an NRS-11 pain score of ≥4. Two hours after IV paracetamol,if the NRS-11 score≥4, 50 mg of tramadol HCL will be administered IV as the second rescue treatment.In addition, when the NRS score is ≥4 at follow-up, paracetamol 1 g, IV will be administered with dosing intervals not shorter than 6 hours.
  Arms: block group
Procedure: parenteral local anesthesia — Only local anesthesia 400 mg(20ml) prilocaine 2% prilocaine to surgical field will be applied to the patients who will be inserted cardiac implantable electronic devices.
  An additional 100 mg of prilocaine will be administered as the first-line rescue treatment if the intraoperative NRS-11 score was ≥4.If the patient has an NRS-11 score of ≥4 again during the procedure,100 mg of prilocaine will be administered again as the second rescue treatment.
  In the postoperative follow-up of the patients,1 g of paracetamol will be administered IV as an infusion for 20 minutes as the first rescue treatment if the patients have an NRS-11 pain score of ≥4. Two hours after IV paracetamol,if the NRS-11 score≥4, 50 mg of tramadol HCL will be administered IV as the second rescue treatment.In addition, when the NRS score is ≥4 at follow-up, paracetamol (1 g, IV) will be administered with dosing intervals not shorter than 6 hours.
  Arms: control group

SUMMARY:
Rhomboid intercostal plane block (RIB) has been described in the last decade. Various clinical applications have been found to provide hemithorax analgesia. The use of cardiac implantable electronic devices (CIEDs) is increasing due to comorbidities in the elderly population. Increased myocardial stress with pain in these patients may increase the frequency of adverse cardiac events. Therefore, perioperative pain management ensures patient welfare, reduces complications, and maintains stable hemodynamic values. In this study, we aimed to evaluate the outcomes of RIB in terms of perioperative analgesia and patient and physician satisfaction in patients undergoing CIED.

DETAILED DESCRIPTION:
In accordance with the study design, a randomization list for the two groups is generated by an independent individual using a computer-assisted program (www.randomizer.org). Equal numbers of participants are assigned to either the intervention or control group in a 1:1 ratio. Patients included in the study will be randomized into two groups of 25 patients each. One group (local anaesthesia group - LAG) will receive only local anaesthesia (prilocaine 2%) as per the standard procedure of the institution. The other group (RIB group - RIBG) will receive RIB in addition to the standard procedure. Demographic and clinical data regarding the patients and the procedures performed will be recorded. Information about the first and second rescue treatments in cases of pain during the procedure, as well as the first and second rescue treatments during postoperative follow-up, will also be documented in the same database. Pain levels during the procedure, at the end of the procedure, and at 3, 6, 12, and 24 hours postoperatively will be assessed using the NRS-11. Patient and physician satisfaction will be evaluated using a five-point Likert scale. This study aims to evaluate the efficacy of RIB in patients undergoing CIED implantation by performing pain assessments with the Numeric Rating Scale-11 (NRS-11) during the procedure and the postoperative period. As a secondary outcome, patient and physician satisfaction levels will be assessed during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* no previous ICD or Pacemaker implantation attempt
* ASA ( American Society of Anesthesiologists ) score of 2-3,
* INR < 2.0 ,
* Signing the volunteer consent form,
* Patients who met the study criteria will be included in the study.

Exclusion Criteria:

* Morbidly obese patients (BMI>35 kg/m2),
* Advanced decompensated heart failure with New York Heart Association (NYHA) stage 4,
* Having severe chronic obstructive pulmonary disease,
* Allergy to the prescribed medications ,
* Those who have a skin infection or lesion in the area to be blocked,
* Cannot be communicated and cannot be given a position,
* Severe psychosis and progressive neurological deficits and muscle disease,
* ICD/ Pacemaker revision or upgrade to be made,
* ICD battery replacement
* Pregnant patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The pain will be assessed by the Numeric Rating Scale-11(NRS -11). Minimum pain score is point zero, maximum pain score is ten points. | 4 months
  to measure the analgesic efficacy of RIB
Investigation patient and physician satisfaction assessed by 5-point Likert scale. One point represents strongly unsatisfied and 5 points represent strongly satisfied. | 4 months
  For patient and physician satisfaction;5-point Likert scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, Study Chair — Proffessor
Locations (1):
- Istanbul Universtiy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No